CLINICAL TRIAL: NCT00288782
Title: Receptor Occupancy Determined by PET Neuroimaging of [11C]Mirtazapine in Healthy Humans
Brief Title: PET Neuroimaging of [11C]Mirtazapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other); Fund for Advancement of Medical Science (Unknown); Max Woerzner's Research Award (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Mirtazapine_Occupancy_01_2005
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Mental Disorders; Mood Disorders; Affective Disorders; Depressive Disorders
Keywords: Mirtazapine; Antidepressant; Positron Emission Tomography
MeSH Terms: conditions — Mental Disorders; Mood Disorders; Depressive Disorder | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mirtazapine

SUMMARY:
Recent studies show that 25 - 30% of depressed patients never fully recover, resulting in a treatment-resistant condition. Thus, depression is a major cause of human suffering. We are interested in finding new ways of identifying and alleviating treatment-resistant depression, and we believe that recent advances in brain imaging can contribute to achieving that goal. In this project, we will use a novel compound ([N-methyl-11C]mirtazapine) that we invented for examining the neurochemistry of brain receptors involved in antidepressant actions.

Our compound, [N-methyl-11C]mirtazapine, is closely related to the clinically effective antidepressant drug mirtazapine (Remeron®). It labels several types of noradrenergic receptors that have often been implicated in "stress reactions" as well as depressive disorders. We believe that our compound can identify specific molecular brain dysfunctions that are causally related to treatment-resistant depression.

The purpose of this study is to determine whether there is a reliable relationship between the level of mirtazapine in the bloodstream and the occupancy of neuroreceptors by mirtazapine in the brain. We will apply our standard procedures of PET brain scanning and region-of-interest data analysis, using healthy volunteers who will receive a daily dose of mirtazapine (double-blind design with placebo, 7.5 mg or 15 mg daily for 5 days). We believe that this project could provide a procedure for assessing brain function in treatment-resistant depression, with the aim of improving the guidelines for successful, evidence-based treatment of depression.

DETAILED DESCRIPTION:
This project uses a double-blind, placebo-controlled, parallel-group design to determine whether there is a reliable relationship between the level of the antidepressant drug mirtazapine in the bloodstream and the degree of occupancy of neuroreceptors in the brain of healthy human volunteers. The primary data endpoints of the study will be the binding potential of C-11 labelled racemic mirtazapine in the brain under baseline conditions and after 5 days of ingestion of either a placebo tablet or a table containing 7.5 mg or 15 mg of mirtazapine. The degree of receptor occupancy obtained during each experimental condition will be calculated on the basis of the binding potentials in brain regions using data obtained by positron emission tomography (PET scanning). Blood samples will be obtained at the time of PET scanning in order to determine whether there is a reliable correlation between the concentration of mirtazapine in the bloodstream and the degree of receptor occupancy achieved in brain. The study plans to include 24 healthy volunteers with 8 subjects in each of the three groups (placebo, 7.5 mg mirtazapine, and 15 mg mirtazapine). Subjects will be randomized into groups in such a way that each of the three treatments will be used for each of three consecutive subjects that enter the study. This procedure will reduce the possibility that differences in procedures that might occur over time will introduce bias into the results. Radiosynthesis of (C-11)mirtazapine will occur by the authorized and documented procedures currently established at the PET Center of Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Drug-free
* No cognitive impairment
* Normal brain anatomy based on MRI
* Contraceptive use by females

Exclusion Criteria:

* PET scanned during past year
* Chronic illness
* Daily use of drug
* Mental illness
* Abnormal value in routine blood analysis
* Pregnancy
* Breast feeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Binding potential in brain regions at tine of each PET scan
Serum concentration at time of each PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Donald F Smith, PhD, DMSc, Principal Investigator — Center for Basic Psychiatric Research, Psychiatric Hospital of Aarhus University, Skovagervej 2, 8240 Risskov, Denmark
Locations (1):
- Center for Psychiatric Research, Psychiatric Hospital of Aarhus University, Risskov, Denmark